CLINICAL TRIAL: NCT01561690
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of ARRY-502 in Adults With Persistent Asthma
Brief Title: A Study of ARRY-502 in Patients With Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARRAY-502-201; C4681001 (Other: Alias Study Number)
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARRY-502 (Experimental)
  Interventions: Drug: ARRY-502, CRTh2 antagonist; oral
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; oral

INTERVENTIONS:
Drug: ARRY-502, CRTh2 antagonist; oral — multiple dose, single schedule
  Arms: ARRY-502
Drug: Placebo; oral — matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2 study, involving a 6-week treatment period, designed to evaluate the effectiveness of investigational study drug ARRY-502 in treating mild to moderate persistent asthma, and to further evaluate the safety of the drug. Approximately 180 patients from the US will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented history of bronchial asthma diagnosed at least 6 months prior to study start and prior to the age of 40 years.
* Body mass index (BMI) of 18 to 35 inclusive.
* An ACQ score of ≥ 1.5 at specified time points prior to first dose of study drug.
* A best prebronchodilator FEV1 of 60% to 85% of the predicted normal value and a change in best postbronchodilator FEV1 of ≥ 12% and ≥ 200 mL at specified time points prior to first dose of study drug.
* Additional criteria exist.

Key Exclusion Criteria:

* Evidence of aspirin-sensitive asthma.
* Pre-existing lung disease other than asthma.
* Clinically significant dermatologic, hematological, renal, endocrine, pulmonary (other than asthma), gastrointestinal, cardiovascular, hepatic, neurologic, ophthalmologic, musculoskeletal or immunologic disease (excepting allergic disease and asthma) that is uncontrolled despite treatment or is likely in the opinion of the Investigator to require a change in therapy during the study.
* Patients with any current or past history of cancer within 5 years prior to study start except for treated basal cell or squamous cell carcinomas of the skin, ductal carcinoma in situ of the breast or cervical carcinomas in situ.
* Any history of serious illness requiring hospitalization within 6 months prior to study start.
* Known positive serology for the human immunodeficiency virus (HIV), hepatitis B and/or active hepatitis C.
* A positive test for drugs or alcohol, unless the positive drug screen is associated with a prescribed medication and is approved by the Medical Monitor.
* Smoking (tobacco or marijuana) within 6 months prior to study start and/or a smoking history of > 10 packs/year.
* Blood donation of ≥ 1 pint (473 mL) within 8 weeks prior to the first dose of study drug.
* Previous treatment with ARRY-502.
* Additional criteria exist.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2012-04-02 (Actual); Primary Completion 2013-05-31 (Actual); Study Completion 2013-06-10 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of the study drug (versus placebo) in terms of prebronchodilator forced expiratory volume in 1 second (FEV1). | 6 weeks

SECONDARY OUTCOMES:
Characterize the safety profile of the study drug in terms of adverse events, clinical laboratory tests, vital signs and electrocardiograms. | 6 weeks
Measure the exposure of study drug in terms of plasma concentrations. | 6 weeks
Assess the effect of study drug on asthma control in terms of Asthma Control Questionnaire (ACQ) score, the number of symptom-free days and the number of weekly short-acting beta (ß) 2 agonist (SABA) metered dose inhaler (MDI) actuations. | 6 weeks
Assess the effect of study drug on respiratory function in terms of FEV1, forced vital capacity (FVC), forced expiratory flow (FEF) and peak expiratory flow (PEF). | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (43):
- United States (43):
  - Allergy & Asthma Specialists Medical Group, Huntington Beach, California
  - Allergy Medical Clinic - Research Division, Los Angeles, California
  - California Allergy & Asthma Med. Group, Los Angeles, California
  - Southern California Institute for Respiratory Diseases Inc, Los Angeles, California
  - Southern California Research, Mission Viejo, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Allergy Associates Medical Group, San Diego, California
  - Colorado Allergy and Asthma Center, Centennial, Colorado
  - IMMUNOe International Research Centers, Centennial, Colorado
  - Asthma & Allergy Associates PC, Colorado Springs, Colorado
  - Rocky Mountain Center for Clinical Research, Wheat Ridge, Colorado
  - Clinical Neuroscience Solutions, Jacksonville, Florida
  - Pulmonary Disease Specialists, Kissimmee, Florida
  - South Florida Research Trials, Miami, Florida
  - Allergy & Asthma Diagnostic Treatment Center, Tallahassee, Florida
  - Florida Pulmonary Research Institute, Winter Park, Florida
  - Idaho Research, Eagle, Idaho
  - Sneeze, Wheeze & Itch, Normal, Illinois
  - Chesapeake Clinical Research Inc, Baltimore, Maryland
  - Northeast Medical Research Associates, North Dartmouth, Massachusetts
  - Clinical Research Institute, Minneapolis, Minnesota
  - Clinical Research Institute, Plymouth, Minnesota
  - Clinical Research Group of Montana, Bozeman, Montana
  - The Asthma & Allergy Center, Bellevue, Nebraska
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Allergy, Respiratory & Sleep Center, Canton, Ohio
  - Bernstein Clinical Research, Cincinnati, Ohio
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Allergy Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Baker Allergy, Asthma & Dermatology Research Center, Lake Oswego, Oregon
  - Clinical Research Institute of Southern Oregon, Medford, Oregon
  - University of Pittsburgh Asthma Institute, Pittsburgh, Pennsylvania
  - Tekton Research, Austin, Texas
  - Pharmaceutical Research & Consulting Inc., Dallas, Texas
  - Western Sky Medical Research Inc, El Paso, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Asthma Inc., Seattle, Washington
  - Allergy Asthma & Sinus Center, S.C., Greenfield, Wisconsin
  - Asthma Allergy & Pulmonary Research, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests